CLINICAL TRIAL: NCT06666322
Title: Platform Trial For Cryptococcal Meningitis
Acronym: PLATFORM-CM
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDIM-2024-32879
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Hiv; Cryptococcal Meningitis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Meningitis, Cryptococcal | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Control group (Active Comparator): randomized to standard of care
  Interventions: Drug: Standard of care
- Experimental group 1 (Experimental): randomized to experimental antifungal therapy #1
  Interventions: Drug: Oteseconazole - antifungal therapy 1
- Experimental group 2 (Experimental): randomized to experimental antifungal therapy #2
  Interventions: Drug: Sfu-AM2-19 Injection - antifungal therapy 2
- Experimental group 3 (Experimental): randomized to experimental antifungal therapy #3
  Interventions: Drug: Antifungal therapy 3
- Experimental group 4 (Experimental): randomized to experimental antifungal therapy #4
  Interventions: Drug: Antifungal therapy 4

INTERVENTIONS:
Drug: Standard of care — 2022 WHO First Line Induction Therapy:
  1. Liposomal Amphotericin B 10mg/kg IV given once
  2. Flucytosine 100mg/kg/day for 14 days in divided doses
  3. Fluconazole 1200mg/day for 14 days Consolidation Therapy: Fluconazole 800mg/day from 2 to 10 weeks Secondary Prophylaxis: Fluconazole 200mg/day through 1 year minimum
  Arms: Control group
Drug: Oteseconazole - antifungal therapy 1 — Oteseconazole, is an azole metalloenzyme inhibitor targeting the fungal sterol, 14α demethylase (CYP51)
  * Loading doses of oral Oteseconazole 600 mg twice daily for 10 days, then 600 mg oteseconazole weekly on weeks 3, 4, 5, and 6.
  * Liposomal Amphotericin B 10 mg/kg IV once.
  * No fluconazole or 5FC to be given.
  Arms: Experimental group 1
Drug: Sfu-AM2-19 Injection - antifungal therapy 2 — SF001 2.0 mg/kg IV administered on day 1, followed by 1.5 mg/kg on day 8 with Fluconazole 1200mg/day and flucytosine 100mg/day in divided doses x 14 days
  Arms: Experimental group 2
Drug: Antifungal therapy 3 — To be determined
  Arms: Experimental group 3
Drug: Antifungal therapy 4 — To be determined
  Arms: Experimental group 4

SUMMARY:
Cryptococcal meningitis is a fungal infection that causes a severe syndrome of meningitis that is 100% fatal without antifungal therapy. Even with antifungal therapy, mortality rates remain high, especially in low and middle income countries where the ongoing HIV/AIDS pandemic increases the risk of cryptococcosis among persons living with HIV infection. The combination of amphotericin and flucytosine (5-FC) has been the mainstay of therapy for the initial management of cryptococcal meningitis for 4 decades. Indeed, the effective delivery of these first line therapy in Africa can lower mortality to 25%. However, several challenges exist. First, even while 5-FC is included on the WHO list of essential medicines, the availability of 5-FC worldwide is limited. Second, liposomal amphotericin (Ambisome ®) is currently available from a single source supplier, creating risk. Third, current therapies have substantial toxicity. Lastly, with widespread agricultural fungicide use of azoles, the median fluconazole minimum inhibitory concentration (MIC50 ) for Cryptococcus has doubled since 2013. Globally, new or improved antifungals are needed for cryptococcal meningitis, particularly those which have less toxicity, greater efficacy, a prolonged half-life, and minimal drug-drug interactions. As multiple new antifungal medicines are on the horizon, this platform trial utilizes a master protocol to investigate, multiple regimens using standardized eligibility criteria, standardized study schedule of events, and standardized contemporary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* CSF cryptococcal antigen (CrAg) positive meningitis
* Living with HIV
* Ability and willingness to provide informed consent
* Willing to receive protocol-specified lumbar punctures
* Age >= 18 years
* Female participants of childbearing potential who are participating in sexual activity that could lead to pregnancy must agree to use reliable forms of contraception (duration will be indicated in each Trial Appendix).

Exclusion Criteria:

* Received 3 or more doses of antifungal therapy for meningitis within last 30 days
* Inability to take enteral (oral or nasogastric) medicine
* Cannot or unlikely to attend regular clinic visits
* Receiving chemotherapy or corticosteroids
* Receiving hemodialysis or known liver cirrhosis
* Suspected Paradoxical immune reconstitution inflammatory syndrome (IRIS)
* Pregnancy or breastfeeding
* Previous administration of investigational study drug
* Any condition for which participation would not be in the best interest of the participant or that could limit protocol specified assessments
* Trial Appendix study-drug specific eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2032-04-21 (Estimated); Study Completion 2032-04-21 (Estimated)

PRIMARY OUTCOMES:
Rate of cerebrospinal fluid (CSF) Cryptococcus clearance (Early Fungicidal Activity, or EFA) | 2 weeks
  quantified by the change of log 10 Cryptococcus CFU/mL CSF/day as measured by serial quantitative CSF fungal cultures over ~2 weeks.
All-cause mortality | 2 weeks
  measured at 2-weeks

SECONDARY OUTCOMES:
Desirability of Outcome Response (DOOR) as ordinal ranked maximum score tested by Win Ratio. | 18 weeks
  1. Death by 18-weeks
  2. Serious Adverse Event through 18 weeks (e.g. all-cause re- hospitalization, permanent neurologic deficit, etc.), lost to follow up before 10-weeks.
  3. Grade 4 lab adverse event by 10 weeks, early discontinuation of study drug, or lost to follow up after 10 weeks.
  4. Grade 3 lab adverse event by 10 weeks OR study drug interruption or dose reduction
  5. Survival through 18-weeks
Survival time through 18 weeks without Cryptococcus culture-positive relapse of meningitis | 18 weeks
  number of participants
CSF culture sterility (cumulative incidence over 18 weeks) | 18 weeks
18-week survival time | 18 weeks
Use of rescue/additional IV amphotericin beyond scheduled use | 18 weeks
Modified Rankin score on functional status at 18 weeks | 18 weeks
Incidence of laboratory abnormalities by Grade 1-5 | 10 weeks
Incidence of serious adverse events | 18 weeks
Incidence of study drug discontinuation or interruption >1 day due to toxicity, by adverse event grade. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David R Boulware, MD, MPH, Principal Investigator — University of Minnesota; David B Meya, MBChB, MMed, PhD, Principal Investigator — Uganda
Locations (2):
- Uganda (2):
  - Infectious Diseases Institute, Kampala
  - Mbarara University of Science and Technology, Mbarara